CLINICAL TRIAL: NCT03931317
Title: A Randomized, Single Center, Masked, Crossover Study Comparing the Effects of Latanoprostene Bunod and Timolol on Retinal Blood Vessel Density and Visual Acuity in Patients With Ocular Hypertension or Primary Open Angle Glaucoma
Brief Title: Study Comparing the Effects of Latanoprostene Bunod and Timolol on Retinal Blood Vessel Density and Visual Acuity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Diego (Other)
Collaborators: Bausch & Lomb Incorporated (Industry)
Responsible Party: Principal Investigator, Robert Weinreb, Distinguished Professor and Chair, Ophthalmology, University of California, San Diego
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: 180658
Record Dates: First submitted 2019-03-31; First posted 2019-04-30 (Actual); Last update posted 2023-08-29 (Actual); Status verified 2023-08

CONDITIONS: OAG - Open-Angle Glaucoma; OHT - Ocular Hypertension
MeSH Terms: conditions — Glaucoma, Open-Angle; Ocular Hypertension | interventions — BOL 303259-X; Timolol; BID protein, human

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Latanoprostene bunod 0.024% QD (Other): 4 weeks of Latanoprostene bunod 0.024% QD, then a 2 Week washout, followed by 4 weeks of Timolol maleate 0.5% BID
  Interventions: Drug: Latanoprostene bunod 0.024% QD
- Timolol maleate 0.5% BID (Other): 4 weeks of Timolol maleate 0.5% BID, then a 2 Week washout, followed by 4 weeks of Latanoprostene bunod 0.024% QD
  Interventions: Drug: Timolol maleate 0.5% BID

INTERVENTIONS:
Drug: Latanoprostene bunod 0.024% QD — This is a randomized, single-center, investigator-masked, 2-period, 8-week treatment study with washout and crossover between treatment periods. There will be 2 treatments in this study: latanoprostene bunod 0.024% QD and timolol maleate 0.5% BID.
  Other Names: Vyzulta
  Arms: Latanoprostene bunod 0.024% QD
Drug: Timolol maleate 0.5% BID — This is a randomized, single-center, investigator-masked, 2-period, 8-week treatment study with washout and crossover between treatment periods. There will be 2 treatments in this study: latanoprostene bunod 0.024% QD and timolol maleate 0.5% BID.
  Other Names: Timoptic
  Arms: Timolol maleate 0.5% BID

SUMMARY:
The purpose of this research study is to compare the effect of Latanoprostene Bunod and Timolol on eye pressure and blood vessels of the back of the eye.

DETAILED DESCRIPTION:
The primary objective of this clinical investigation is to compare the difference in change in retinal blood vessel density (peripapillary and macular) between latanoprostene bunod (LBN) ophthalmic solution 0.024% dosed once daily (QD) and timolol maleate 0.5% dosed twice daily (BID) in subjects with OAG or OHT and in normal subjects.

Primary Efficacy Endpoint The primary efficacy endpoint for this study is the change in retinal blood vessel density (peripapillary and macular) between treatment groups after 4 weeks of treatment (Visit 4 [Week 5] and Visit 6 [Week 11]).

Secondary Efficacy Endpoints The secondary efficacy endpoint for this study is change in best-corrected visual acuity (BCVA).

Safety Endpoints The safety endpoint for this study is the incidence of ocular and systemic adverse events (AEs).

ELIGIBILITY:
Inclusion Criteria:

* Subjects must be between 40 to 90 years of age, inclusive, on the date the Informed Consent Form (ICF) is signed and with the capacity to provide voluntary informed consent.
* Subjects must be able to read, understand, and provide written informed consent on the Institutional Review Board (IRB) approved ICF. Only English speakers will be enrolled.
* Subjects who are able and willing to comply with all treatment and follow-up/study procedures.
* Female subjects who are not of childbearing potential or female subjects who have a negative urine pregnancy test result at Visit 1 (Screening) and Visit 3 (Randomization, Week 1).
* Females of childbearing potential, defined as a female who is fertile following menarche, must have a negative serum pregnancy test at screening and agree to use an acceptable method of contraception throughout their participation in the study.

Exclusion Criteria:

* Subjects participating in any drug or device clinical investigation within 30 days prior to Visit 1 (Screening) for subjects requiring a washout period, or 30 days prior to Visit 3 (Randomization, Week 1) for treatment naïve subjects.
* Subjects who anticipate participating in any other drug or device clinical investigation within the duration of this study.
* Subjects with a history or presence of chronic generalized systemic disease that the Investigator feels might increase the risk to the subject or confound the results of the study.
* Female subjects who are pregnant or breastfeeding.
* Subjects currently taking systemic β-adrenergic antagonists.
* Subjects with an anticipated need to initiate or modify medication (systemic or topical) that is known to affect IOP (eg, α-adrenergic agonists, calcium channel blockers, angiotensin converting enzyme [ACE] inhibitors, and angiotensin II receptor blockers).
* Subjects with known hypersensitivity or contraindications to latanoprostene bunod or any of the ingredients in the study drugs.
* Subjects with known hypersensitivity or contraindications to timolol maleate or other -adrenergic receptor antagonists or any of the ingredients in the study drugs.
* Subjects who are expected to require treatment with ocular or systemic corticosteroids.
* Subjects who are in need of any other topical or systemic treatment of OAG or OHT.
* Subjects who are unable to discontinue contact lens use during and for 15 minutes following instillation of study drug and for 24 hours before check-in to and during each study visit.
* Subjects with a central corneal thickness greater than 600 µm in either eye, measured by pachymetry.
* Subjects with any condition that prevents reliable applanation tonometry (eg, significant corneal surface abnormalities) in either eye.
* Subjects with advanced glaucoma.
* Subjects with any condition that prevents clear visualization of the fundus in either eye.
* Subjects who are monocular.
* Subjects with previous or active corneal disease in either eye.
* Subjects with current or a history of severe dry eye in either eye.
* Subjects with active optic disc hemorrhage in either eye.
* Subjects with current or a history of central/branch retinal vein or artery occlusion in either eye.
* Subjects with current or a history of macular edema in either eye.
* Subjects with very narrow angles (3 quadrants with less than Grade 2 according to Shaffer's anterior chamber angle grading system) and subjects with angle closure, congenital, and secondary glaucoma, and subjects with history of angle closure in either eye.
* Subjects with a diagnosis of a clinically significant or progressive retinal disease (eg, diabetic retinopathy, macular degeneration) in either eye.
* Subjects with any intraocular infection or inflammation in either eye within 3 months prior to Visit 1 (Screening).
* Subjects with a history of ocular laser surgery in either eye within the 3 months prior to Visit 1 (Screening).
* Subjects with a history of incisional ocular surgery or severe trauma in either eye within 3 months prior to Visit 1 (Screening).

Ages: 40 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2018-12-03 (Actual); Primary Completion 2021-05-20 (Actual); Study Completion 2023-03-01 (Actual)

PRIMARY OUTCOMES:
retinal blood vessel density (peripapillary and macular) | Through study completion, an average of 11 to 19 weeks
  The primary efficacy endpoint for this study is the change in retinal blood vessel density (peripapillary and macular) between treatment groups after 4 weeks of treatment (Visit 4 [Week 5] and Visit 6 [Week 11]).

SECONDARY OUTCOMES:
best-corrected visual acuity (BCVA) | Through study completion, an average of 11 to 19 weeks
  The secondary efficacy endpoint for this study is change in best-corrected visual acuity (BCVA)

OTHER OUTCOMES:
Safety Endpoints: incidence of ocular and systemic adverse events (AEs) | Through study completion, an average of 11 to 19 weeks
  The safety endpoint for this study is the incidence of ocular and systemic adverse events (AEs)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Weinreb, MD, Principal Investigator — UCSD Shiley Eye Institute
Locations (1):
- UCSD Shiley Eye Institute, La Jolla, California, United States